CLINICAL TRIAL: NCT02298738
Title: Relation of Low Vitamin D Levels and New-onset AF Among Hypertensive Patients
Brief Title: Effect of Vit D on New-onset AF in Hypertension
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Özgür Ulaş Özcan, Dr Ozgur Ulas Ozcan, Ankara University
Other Study IDs: AnkaraU
Record Dates: First submitted 2014-11-20; First posted 2014-11-24 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Atrial Fibrillation; Hypertension
Keywords: Atrial fibrillation, hypertension, vitamin D
MeSH Terms: conditions — Atrial Fibrillation; Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- New onset Atrial fibrillation: New-onset AF was defined as patients with hypertension and atrial fibrillation which was identified for the first time by an electrocardiogram or ambulatory holter monitoring.
- control: Hypertensive patients without atrial fibrillation.

SUMMARY:
Atrial fibrillation (AF), an important cause of cardiac mortality and morbidity is the most common type of cardiac arrhythmia in clinical practice. Hypertensive individuals are at particular risk of development of atrial fibrillation. Renin-angiotensin-aldosteron system (RAS) which is activated in hypertension may be the underlying mechanism of AF among hypertensive patients.

Vitamin D deficiency has been shown to be involved in the pathogenesis of hypertension, cardiovascular disease and obesity. Increased RAS activity is one of the postulated mechanisms by which vitamin D deficiency may trigger the development of hypertension and various cardiovascular diseases. On the basis of these data we hypothesized that hypovitaminosis D might be associated with new-onset AF among patients with hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patients with new-onset AF

Exclusion Criteria:

Established coronary artery disease

* Heart failure
* Chronic obstructive pulmonary disease
* Diabetes mellitus
* Significant heart valve disease
* Hyperthyroidism
* Renal failure
* Any malignancy
* Acute infection
* Recent thoracic or abdominal surgery
* Under therapy of Vit D3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertensive patients with new-onset AF. New onset AF was defined as AF identified for the first time by an electrocardiogram or ambulatory holter monitoring. Hypertension was defined as blood pressure ≥ 140/90 mmHg or a history of antihypertensive drug use.
Sampling Method: Non-Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2012-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
hypovitaminosis D | Baseline
  Identifying whether hypovitaminosis D is a risk factor for development of new-onset AF among hypertensive patients